CLINICAL TRIAL: NCT05622032
Title: Blood Virome After Haploidentical Hematopoietic Stem Cell Transplantation, a Pilot Study
Status: Completed | Type: Observational
Sponsor: Laurent Kaiser (Other)
Responsible Party: Sponsor-Investigator, Laurent Kaiser, Head, Division of Infectious Diseases, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: Blood virome after haplo-HSCT
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Haploidentical Hematopoietic Stem Cell Transplantation
Keywords: viral infection; blood virome
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood specimens originating from the above biobank, collected at 4 time points (day 0, 30, 90 and 180) after transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- haploidentical HSCT patients: Patients receiving HSCT from a haploidentical donor. They also receive a treatment called cyclophosphamide as part of the protocol to prevent graft versus host disease at day 3 and 4 after transplantation.
- HLA-matched HSCT patients: Patients who receive HSCT from a HLA-matched donor.

SUMMARY:
The goal of this observational study is to assess the risk of viral infections in patients receiving hematopoietic stem cell transplantation (HSCT) from a haploidentical donor compared to those who receive HSCT from a HLA-matched donor. The main question it aims to answer is: to describe which viruses are replicating in the blood of the above two patient groups on the day of transplantation and at 1, 3 and 6 months after transplantation. Blood samples taken as part of routine care on the day of transplantation and at 1, 3 and 6 months post-transplantation visits are analyzed and the types and amount of viruses detected in the two groups of patients are described.

DETAILED DESCRIPTION:
Geneva University Hospitals are one of the three centers performing allogeneic HSCT in Switzerland. Since several years the Division of infectious diseases runs a collaborative research program with the Division of Hematology. In 2015 the two divisions jointly created a prospective cohort of allo-HSCT patients called: "Infectious diseases in hematopoietic stem cell transplant patients cohort" enrolling potentially all adult patients engrafted in our center since 2015 (CCER protocol 15-120 and relative amendments). The cohort compiles clinical data on hematological and infectious complications occurring up to one year after transplantation and biological specimen collected systematically until up to 2 years after transplantation, which are stored in a joint biobank.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving allogeneic stem cell transplantation at the Geneva University Hospitals from a haploidentical or from an HLA-matched donor, who signed the informed consent form before transplantation for inclusion in the prospective cohort of "Infectious disease in hematopoietic stem cell transplant patients".

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving allogeneic HSCT at the Geneva University Hospitals from a haploidentical or from an HLA-matched donor, who signed the informed consent form before transplantation for inclusion in the prospective cohort of "Infectious disease in hematopoietic stem cell transplant patients".
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Describe the blood virome in haploidentical and HLA-matched allo-HSCT recipients during the first 6 months after transplantation. | 6 months after transplantation
  Describe the types of viruses detected as well as their frequency in the blood virome of haplo- HSCT patients compared to the HLA-matched group by metagenomic next generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Kaiser, Pr, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Datasets originating from our project and used in case of the publication of our results will be deposited on the institutional open access data repository: Yareta and will be made public at the time of the publication. Metadata will be searchable and discoverable. Concerning the mNGS data, in case of scientific publication, raw data will be deposited in the publicly available repository Sequence Read Archive (SRA) from NCBI.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the publication of the results
Access Criteria: open access